CLINICAL TRIAL: NCT02426463
Title: Individualising Drug Therapy in Neonates Using Pharmacogenomic Profiling, Population Based Modeling and Simulations
Brief Title: Clinical Trial on Individual Characteristics Affecting Pain Drug Therapy in Neonates
Acronym: NeoPopGen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other); University of Helsinki (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T65/2015
Record Dates: First submitted 2015-04-13; First posted 2015-04-27 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Critical Illness
Keywords: Neonatal intensive care; need for intratracheal intubation
MeSH Terms: conditions — Critical Illness | interventions — Propofol; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol (Active Comparator): Plasma samples and patient data are collected prospectively from 40 neonates who receive propofol as part of their care in the neonatal intensive care unit at the Turku University Hospital, Turku, Finland.
  Interventions: Drug: propofol
- Oxycodone (Active Comparator): Plasma samples and patient data are collected prospectively from 40 neonates who receive oxycodone as part of their care in the neonatal intensive care unit at the Turku University Hospital, Turku, Finland.
  Interventions: Drug: oxycodone

INTERVENTIONS:
Drug: propofol
  Arms: Propofol
Drug: oxycodone
  Arms: Oxycodone

SUMMARY:
Children differ from adults with respect to growth and development but also immaturity of various pharmacological mechanisms. Dosing schemes in children are usually derived in an empirical manner from clinical trials in adult patient groups. All this poses neonates to an increased risk for therapeutic failure and adverse drug reactions.

Medicinal products studied during this project are among the ones with the highest needs for research in the pediatric intensive care. This project focuses on the necessity to integrate subject's individual characteristics to assist clinical decision-making in drug therapy. The investigators explore the mechanisms defining the dose response in pediatric populations. The results obtained with these studies will help to find safer drug dosing regimens in this delicate patient population.

ELIGIBILITY:
Inclusion Criteria:

* Given informed consent by the guardian of an eligible patient.
* Patient is more than 24 weeks old and has a body weight more than 500 g.
* Patient needs intensive care treatment based on a clinical decision by a neonatologist and receives propofol or oxycodone on their therapy. Attending neonatologist makes the decision to prescribe propofol for scheduled short procedural sedation or oxycodone for analgesia as well as all other treatment related decisions.

Exclusion Criteria:

* Eligible patients guardian declines to give informed consent.
* A previous history of intolerance to the study drugs or to related compounds and additives.
* History of any kind of drug allergy.
* Participation in any other studies concomitantly or within one month prior to the entry into this study.

Ages: 24 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2015-04-20 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of propofol and oxycodone. | 24 hours post-dose.
  Primary outcome is to build up a population pharmacometric model to describe pharmacokinetics of propofol and oxycodone based on drug concentrations analyzed from the plasma samples.

SECONDARY OUTCOMES:
Effect of biometric and genomic covariates on AUC | 24 hours post-dose
  Covariate analysis and simulations to individualize population models
Efficacy of propofol in procedural anesthesia in neonates | 24 hours
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability during procedural anesthesia for intratracheal intubation in neonates
Efficacy of oxycodone as an analgesic in neonates during mechanical ventilation | 24 hours
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability in neonates after oxycodone administration during mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Teijo I Saari, MD, PhD, Principal Investigator — Dept. Anaesthesiology and Intensive Care, University Of Turku
Locations (1):
- Department of Paediatrics and Adolescent Medicine, Turku University Hospital, Turku, Finland